CLINICAL TRIAL: NCT00770679
Title: Effects of Statins on Lower Extremity Arterial Function Assessed by Magnetic Resonance Imaging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed recruitment, funding exhausted
Sponsor: Johns Hopkins University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA00002253
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High-Dose Statin (Experimental): 80 mg atorvastatin daily for 3 weeks
  Interventions: Drug: lipitor

INTERVENTIONS:
Drug: lipitor — 80 mg everyday (QD) for 3 weeks
  Other Names: atorvastatin

SUMMARY:
Cholesterol-lowering drugs called statins improve the functioning of the endothelium, and help prevent heart disease. The investigators are testing whether statins improve endothelial function more in the arteries that have worse endothelium to begin with. One of the functions of the endothelium is to help control how blood vessels dilate (expand) or contract (narrow) in different situations. This affects how blood flows through those vessels. Magnetic resonance imaging (MRI) can be used to evaluate endothelial function in the arms and legs noninvasively.

DETAILED DESCRIPTION:
Correct

ELIGIBILITY:
Inclusion Criteria:

* Age 40-90
* Male or female
* Type 2 diabetes

Exclusion Criteria:

* Known pregnancy or nursing.
* Females of child bearing potential must have been surgically sterilized or be post menopausal.
* Smoking
* Known vascular disease
* Inability to complete MRI scan
* Symptoms of claudication
* Use of a nitrate medicine
* Use of any cholesterol-lowering agent
* LDL < 70
* Acute illness
* Liver disease
* Contraindication to getting an MRI scan (i.e. electronic implant, shrapnel, cerebral aneurysm clip, welding history).

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Silber, MD, Principal Investigator — JHU
Locations (1):
- Harry SIlber, MD, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Dose Statin
Started | 16
Completed | 10
Not Completed | 6
Not completed — Lost to Follow-up | 3
Not completed — Follow-up LDL measurement not collected | 3

BASELINE CHARACTERISTICS:
Arm/Group | High-Dose Statin
Number analyzed (Participants) | 16
Age, Customized [Count of Participants; unit: Participants]
  >=40, <=90, years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Low Density Lipoprotein (LDL)
Description: Serum LDL, mg/dL (baseline LDL-follow-up LDL)
Time Frame: Change from baseline to follow-up, up to 5 weeks
Population: 3 participants were lost to follow-up, 3 participants did not have LDL values collected/reported at follow-up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | High-Dose Statin
Number analyzed (Participants) | 10
mg/dL | 75.54 (12.98)

2. Primary Outcome: Change in Endothelial Function as Measured on MRI in the Arms
Time Frame: chance from baseline to end of study, up to 5 weeks
Population: No data was collected for this outcome measure. The outcome was not able to be calculated based upon data obtained and programs and investigator capabilities.
Arm/Group | High-Dose Statin
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Endothelial Function as Measured on MRI in the Legs
Time Frame: chance from baseline to end of study, up to 5 weeks
Population: as for outcome 2
Arm/Group | High-Dose Statin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | High-Dose Statin
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes